CLINICAL TRIAL: NCT06156436
Title: A Study Evaluating the Use of ResAppDx v2.0 as an Aid to Diagnose Respiratory Disease in Paediatric Patients in an Emergency Department
Status: Completed | Type: Observational
Sponsor: ResApp Health Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: 19002
Record Dates: First submitted 2023-11-26; First posted 2023-12-05 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Croup; Bronchiolitis; Asthma in Children; Reactive Airway Disease; Pneumonia; Lower Respiratory Tract Infection
MeSH Terms: conditions — Croup; Bronchiolitis; Pulmonary Disease, Chronic Obstructive; Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Paediatric Patients
  Interventions: Device: ResAppDx v.20

INTERVENTIONS:
Device: ResAppDx v.20 — Software application used to aid diagnosis of respiratory disorders

SUMMARY:
Aim of study is to demonstrate that the ResAppDx v2.0 algorithms provide an accurate diagnosis of paediatric respiratory disease in the study's clinical setting compared to a Clinical Adjudication Committee's (CAC) diagnosis; and to establish a baseline for the resource use and cost of current care pathways for paediatric respiratory disease diagnosis in an emergency department. Eligible subjects/parents will be assented/consented, enrolled and their subject reported signs/symptoms of respiratory disease will be recorded in the study electronic case report form (eCRF).The enrolled subject's cough sounds will be captured (5 cough sounds are required) using the ResAppDx v2.0 Investigational Device (ID) software installed on a study smartphone; cough sounds may be voluntary and/or involuntary/spontaneous. As this is an observational study the treating team will be blinded to the ResAppDx v2.0diagnoses. Additional medical information will be collected from the treating team, from the subject/parent and from the subject's medical record. No follow-up/subsequent visits with the subject will be required by the study. As an efficacy comparator, a CAC will determine the final clinical diagnosis for each enrolled subject using the disease case definitions, eCRF data, the subject's medical record and cough sound recordings.Information on time and scope of tests and consults ordered by the treating team will be recorded to set a baseline for resource use and cost and time of current standard of care treatment/assessment procedures. This data will allow future health economics analyses to be performed.The blinded ResAppDx v2.0diagnoses will be unblinded after database lock and sensitivity and specificity will be calculated for the ResAppDx v2.0diagnoses compared to agreement with the CAC's final clinical diagnoses for this cohort.

ELIGIBILITY:
Inclusion Criteria:

* Infants and children, aged from 29 days to less than 12 years of age.

  1. Presenting to the study site with current signs or symptoms of rhinorrhea, cough, wheeze, stridor, increased work of breathing, cyanosis, additional auscultatory noises (crepitations), or low oximetry levels.
  2. Onset of symptoms must have occurred within the past 14 days.

Exclusion Criteria:

1. Parent or legal guardian is unwilling or unable to sign the study informed consent form.
2. A child who, in the opinion of the investigator, is able to provide assent based on their age, maturity or psychological state is unwilling or unable to sign the study assent form.
3. Patient requires mechanical ventilatory support (including invasive, CPAP, or BiPAP) or high flow nasal cannula
4. Patient has a history of structural airways abnormalities, tracheobronchomalacia, or vocal cord abnormalities (e.g. laryngomalacia, tracheomalacia, or bronchomalacia)
5. Patient has a medical contraindication to voluntary cough, including the following (only enroll if coughing spontaneously)

   * Severe respiratory distress
   * History of pneumothorax
   * Eye, chest, or abdominal surgery in past 3 months
   * Hemoptysis in the past month
6. Patient is too medically unstable to participate in study per treating clinician
7. Patient has a tracheostomy present or tube placed
8. Patient is unable to provide at 5 coughs (voluntary and/or spontaneous)

Ages: 29 Days to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Subjects aged from 29 days to less than 12 years of age presenting to a study site with signs or symptoms of respiratory disease including rhinorrhea, cough, wheeze, stridor, work of breathing, cyanosis, additional auscultatory noises (crepitations), chest in-drawing/retractions or fast breathing.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Efficacy of ResAppDx v2.0 compared to clinical adjudication panel | 6 months
  Efficacy will be compared to the diagnosis formed by consensus of the Clinical Adjudication Committee (CAC) and evaluated using sensitivity and specificity of ResAppDx v2.0 algorithms ("Index Test") to diagnose and rule out the following conditions:
  * croup;
  * bronchiolitis (for patients less than 2 years old only);
  * asthma / reactive airway disease (RAD);
  * pneumonia and
  * lower respiratory tract disease (LRTD)

CONTACTS AND LOCATIONS:
Locations (5):
- United Kingdom (5):
  - Birmingham Children's Hospital, Birmingham
  - Bristol Royal Hospital of Children, Bristol
  - Leicester Royal Infirmary, Leicester
  - Evelina London Children's Hospital, London
  - The Royal London Hospital, London

IPD SHARING:
Plan to Share IPD: No